CLINICAL TRIAL: NCT06710665
Title: Tumor Regression Grade As Predictor of Adjuvant Therapy Benefits in Patients with Esophageal Squamous Cell Carcinoma After Neoadjuvant Therapy
Brief Title: Tumor Regression Grade As Predictor of Adjuvant Therapy
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Collaborators: The First Affiliated Hospital of Xiamen University (Other); Quanzhou First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TRGAT
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Good responders: Good responders (TRG 0-1). The pathologic report of the patient after neoadjuvant combined surgery
  Interventions: Drug: Chemotherapy
- Poor responders: Poor responders (TRG 2-3). The pathologic report of the patient after neoadjuvant combined surgery
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Chemotherapy

SUMMARY:
Neoadjuvant therapy followed by surgery is preferred for locally advanced esophageal squamous cell carcinoma, but the necessity of adjuvant therapy remains controversial. Tumor regression grade reflects the response to neoadjuvant therapy and may predict patient prognosis, yet its role in guiding adjuvant therapy remains unexplored.

DETAILED DESCRIPTION:
We aim to explore the role of TRG and other clinical characteristics in predicting the efficacy of postoperative adjuvant therapy in ESCC patients receiving neoadjuvant therapy. This study Includes patients who underwent R0 esophagectomy for thoracic ESCC after neoadjuvant therapy. Patients will be assessed by TRG and divided into good responders (TRG 0-1) and poor responders (TRG 2-3). The main variable of interest is adjuvant therapy, and the primary outcome is OS, defined as time from diagnosis until death. Cox proportional hazards regression models will be used to calculate hazard ratios and 95% confidence intervals to assess the impact of various variables on survival time.

ELIGIBILITY:
Inclusion Criteria:

(I) underwent R0 resection with either two-field or three-field lymphadenectomy (II) received neoadjuvant therapy such as preoperative radiotherapy, chemoradiotherapy, or combined immunotherapy (III) had esophageal squamous cell carcinoma pathology.

Exclusion Criteria:

(I) Patients with incomplete clinical data or follow-up information (II) Diagnosed with multiple primary malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes patients who underwent R0 esophagectomy for thoracic ESCC after neoadjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | for patients surviving at least 90 days after surgery
  time from diagnosis until death

CONTACTS AND LOCATIONS:
Overall Officials: Bin Zheng, Study Director — Key Laboratory of Cardio-Thoracic Surgery, Fujian Medical University, Fujian Province University, Fu
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No